CLINICAL TRIAL: NCT02197637
Title: Phase II Trial of Oral Vinorelbine in Children With Recurrent or Progressive Unresectable Low-Grade Glioma
Acronym: OVIMA-1210
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Oscar Lambret (Other)
Collaborators: National Cancer Institute, France (Other Government); Pierre Fabre Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OVIMA-1210; 2013-001625-12 (EudraCT Number); PHRC 12- 194 (Other Grant/Funding Number: INCA)
Record Dates: First submitted 2014-05-09; First posted 2014-07-23 (Estimated); Last update posted 2020-11-18 (Actual); Status verified 2020-11

CONDITIONS: Low-Grade Glioma
MeSH Terms: interventions — Vinorelbine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ORAL VINORELBINE (Experimental): Orally vinorelbine 60 mg/m2 D1, 8 and 15 Cycle of 28 days For a maximum of 12 cycles The dose of vinorelbine should be increased to 80 mg/m2 from the 2nd cycle
  Interventions: Drug: ORAL VINORELBINE

INTERVENTIONS:
Drug: ORAL VINORELBINE — Orally vinorelbine 60 mg/m2 D1, 8 and 15 Cycle of 28 days For a maximum of 12 cycles The dose of vinorelbine should be increased to 80 mg/m2 from the 2nd cycle If on D8 and D15, the administration conditions are not met, the administration is canceled and not delayed.
  Other Names: NAVELBINE

SUMMARY:
The purpose of this study is to determine whether oral vinorelbine is effective in the treatment of children with progressive or recurrent unresectable low grade glioma.

DETAILED DESCRIPTION:
The aim of this study is to determine efficacy of oral vinorelbine in children with progressive or recurrent unresectable low grade glioma, in addition to safety, pharmacokinetic, pharmacogenetic, medical costs and quality of life.

ELIGIBILITY:
Inclusion Criteria:

TUMOR CHARACTERISTICS:

* Histologically confirmed recurrent or progressive primary Low-Grade Glioma (LGG) defined as follow (WHO classification 2007): optic pathway glioma (OPG), pilocytic astrocytoma (PA), fibrillary or diffuse astrocytoma (DA), oligodendroglioma (OG) or oligoastrocytoma (OA)
* Patients with OPG do not require biopsy confirmation of disease, if clinical and radiological findings as well as ophthalmological examination are unequivocal
* Low-Grade Glioma involving the brainstem can be included in case of histological confirmation
* Tumor has to be considered as non totally resectable

PATIENT CHARACTERISTICS:

* Age 6-18 years old
* Lansky or Karnofsky status more than 50 %
* Measurable disease on cerebral and/or spinal MRI, with at least 1 lesion diameter superior to 1 cm
* Patients with metastatic disease are eligible, but at least 1 lesion must be measurable as previously defined
* Patients must have received at least 1 prior chemotherapy regimen containing carboplatin
* Life expectancy of at least 3 months
* Evidence of adequate organ functions, including:
* neutrophil count (ANC) ≥ 1500/mm3 ,
* platelet count ≥100 000/mm3 ;
* serum creatinine < 1.5 x normal for age when the serum creatinine is ≥ 1.5 × the ULN, the glomerular filtration rate (either estimated or formal) must be > 70 mL/min/1.73m2;
* total bilirubin< 1.5 x normal for age,
* ASAT and ALAT < 2.5 x normal for age
* Effective contraception for patients (male and female) with reproductive potential, and for a minimum of 3 months after the end of treatment
* Negative pregnancy test, if applicable
* Patients able to swallow capsules
* Patient affiliated with a health insurance system
* Written informed consent of patient and/or parents/guardians prior to the study participation.

PRIOR OR CONCURRENT THERAPY

* Prior treatments containing vinca alkaloids like vincristine and/or vinblastine are authorized
* Patients must have fully recovered from the toxic effects of any prior therapy before entering the study. No organ toxicity superior to grade 2 according to NCI-CTCAE v4.0
* An interval of at least 2 months from prior radiotherapy, 6 weeks from nitrosourea chemotherapy, and 4 weeks from other chemotherapy regimen, is required

Exclusion Criteria:

* Inclusion criteria failure
* Prior treatment with intravenous or oral vinorelbine
* Known hypersensibility to other vinca-alkaloïdes
* Digestive pathology affecting absorption in a important way
* Prior surgical resection of stomach or the small intestine
* Severe hepatic failure independent from tumoral disease
* Fructose intolerance
* Leptomeningeal relapse without any available measurable disease on MRI (for example, leptomeningeal relapse with totally resected primary lesion)
* Uncontrolled active infection within 2 weeks
* Pregnancy or breast feeding woman
* Uncontrolled intercurrent illness or active infection
* Unsuitable for medical follow-up (geographic, social or mental reasons)
* Patients requiring long-term oxygen therapy
* Patients with ANC less than 1500/mm3
* Patients vaccinated against yellow fever

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 39 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2019-08 (Actual); Study Completion 2020-10 (Actual)

PRIMARY OUTCOMES:
Progression free survival | 9 months
  no progressive disease according to RANO criteria

SECONDARY OUTCOMES:
Response rate | 6 months
  Complete, partial and minor responses according to RANO criteria
Response rate | 12 months
  Complete, partial and minor responses according to RANO criteria
Progression Free Survival PFS | 36 months
  No progressive disease according to RANO criteria
Overall Survival OS | 36 months
  Death incidence
Growth Modulation Index GMI | 36 months
  GMI defined as PFS2/ PSF1 ratio (PFS2 = PFS since the beginning of study treatment ; PFS1 = PFS observed in previous line of treatment)
Adverse events | 12 months
  According to NCI-CTC AE scale v4.0
Modifications of tumor aspects in diffusion and perfusion MRI | At each tumor assessment, after 3, 6, 9 and 12 cycles of treatment, at the end of study, then every 4 months during the first year post therapy, then every 6 months for 3 years, if no prior progressive disease
  Cerebral and/or spinal MRI (morphological and functional) with 2 dimensional assessment of target lesions.
Constitutional polymorphisms of cyp3A5, ABCB1 | Before the start of treatment
  Single nucleotide polymorphisms (SNPs) will be analyzed by real time PCR and correlated with efficacy and toxicity of vinorelbine
Pharmacokinetic | cycles 1 and 2, prior to the initial dose, 30 min, 1, 1.5, 2, 3, 6, 8, 10 and 26 hours post-dose
  Plasmatic concentrations measured by LC-MS/MS (liquid chromatography tandem mass spectrometry) ; Area under the curve (AUC), maximal concentration (Cmax), time to Cmax (Tmax).
Medical costs | during all the study (up to 1 year)
  Costs of medical care including : hospitalisations, emergency admissions, nursing care at home, medical consultations, diet support...
Health Utilities Index (HUI) | Before the treatment, then at day 1 of 1st cycle, after the 3th, 6th, 9th and the 12th cycles of study treatment, and at the end of study (up to 1 year)
  Health Utilities Index (HUI)

CONTACTS AND LOCATIONS:
Overall Officials: Pierre LEBLOND, MD, PhD, Principal Investigator — Centre Oscar Lambret, Lille, France; Nicolas ANDRE, MD, PhD, Principal Investigator — Hôpital La Timone, Marseille, France
Locations (16):
- France (16):
  - CHU d'Angers, Angers
  - CHU de Bordeaux, Bordeaux
  - CHU de Grenoble, Grenoble
  - Centre Oscar Lambret, Lille
  - CHU de Limoges, Limoges
  - Centre Léon Bérard, Lyon
  - Hôpital de la TIMONE, Marseille
  - CHRU Arnaud de Villeneuve, Montpellier
  - CHU de Nancy, Nancy
  - Institut Curie, Paris
  - CHU de Reims, Reims
  - CHU de Rennes - Hôpital Sud, Rennes
  - CHU de Rouen, Rouen
  - Hôpital Hautepierre, Strasbourg
  - Hôpital des Enfants, Toulouse
  - Institut Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: No